CLINICAL TRIAL: NCT01370031
Title: Pilot, Open-Label, Randomized, Repeated Dose, 4-Way Cross-Over, Clinical Pharmacology Study of Beclomethasone Dipropionate (Clenil® Modulite®) 250 µg HFA pMDI Using the Aerochamber Plus™ Spacer Device Versus the Volumatic™ Spacer Device Without or With Charcoal Block in Asthmatic Adults Patients
Brief Title: Pilot Pharmacokinetic Clenil Study With AeroChamber Plus™ or Volumatic™ Spacer Devices
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-1008-PR-0049; 2010-022615-19 (EudraCT Number)
Record Dates: First submitted 2011-04-28; First posted 2011-06-09 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; PK; Adults
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Clenil® Modulite® via AeroChamber Plus™ (Experimental): Clenil® Modulite® administered via AeroChamber Plus™ spacer
  Interventions: Drug: Clenil® Modulite® via AeroChamber Plus™
- Clenil® Modulite® via Volumatic™ (Active Comparator): Clenil® Modulite® administered via Volumatic™ spacer
  Interventions: Drug: Clenil® Modulite® via Volumatic™ spacer
- Clenil® Modulite® via AeroChamber Plus™ plus charcoal block (Experimental): Clenil® Modulite® administered via AeroChamber Plus™ spacer plus charcoal block
  Interventions: Drug: Clenil® Modulite® via AeroChamber Plus™ plus charcoal block
- Clenil® Modulite® via Volumatic™ plus charcoal block (Active Comparator): Clenil® Modulite® administered via Volumatic™ spacer plus charcoal block
  Interventions: Drug: Clenil® Modulite® administered via Volumatic™ spacer plus charcoal block

INTERVENTIONS:
Drug: Clenil® Modulite® via AeroChamber Plus™ — Clenil® Modulite® 250 µg via AeroChamber Plus™ spacer during 14 days
  Arms: Clenil® Modulite® via AeroChamber Plus™
Drug: Clenil® Modulite® via Volumatic™ spacer — Clenil® Modulite® 250 µg via Volumatic™ spacer during 14 days
  Arms: Clenil® Modulite® via Volumatic™
Drug: Clenil® Modulite® via AeroChamber Plus™ plus charcoal block — Clenil® Modulite® via AeroChamber Plus™ spacer during 14 days (plus charcoal block at Day 14)
  Arms: Clenil® Modulite® via AeroChamber Plus™ plus charcoal block
Drug: Clenil® Modulite® administered via Volumatic™ spacer plus charcoal block — Clenil® Modulite® administered via Volumatic™ spacer during 14 days (plus charcoal block at day 14)
  Arms: Clenil® Modulite® via Volumatic™ plus charcoal block

SUMMARY:
The purpose of this study is to evaluate, at steady-state, the systemic exposure and the lung deposition of B17MP (active metabolite of BDP) as AUC0-12h,ss and Cmax,ss, after inhalation of BDP (Clenil® Modulite®) with the AeroChamber Plus™ spacer device or with the Volumatic™ spacer device without or with charcoal block.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female patients aged 18-65 years included.
* Diagnosis of asthma according to GINA guidelines 2009 made at least 6 months prior to screening.
* Patients already treated with a dose of BDP or equivalent up to 2000 µg/day.
* FEV1 ≥ 60% of predicted for the patient's normal value at screening and randomisation

Exclusion Criteria:

* Patients treated with oral or parenteral corticosteroids in the previous 8 weeks (12 weeks for parenteral depot corticosteroids) before screening visit.
* Exacerbation of asthma symptoms or hospitalization due to asthma exacerbation within the previous one month before screening until randomisation.
* Lower respiratory tract infection within one month prior to screening.
* Diagnosis of COPD as defined by the current GOLD 2009 (Global Initiative for Chronic Obstructive Lung Disease) Guidelines.
* Significant medical history and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any laboratory abnormality indicative of a significant underlying condition, that may interfere with patient's safety, compliance, or study evaluations, according to the Investigator's opinion.
* Treatment with a xanthine derivative (e.g. theophylline) formulation in the 4 weeks prior to screening.
* Any enzyme inducing or inhibiting drug (from 8 weeks before screening visit)
* Patients who received any investigational new drug within the last 8 weeks before the screening. The patients cannot participate in another clinical study at the same time as the present study.
* Blood donation (450 mL or more)or significant blood loss less than 12 weeks before the first intake of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Systemic exposure to B17MP (active metabolite of BDP) at steady state after repeated dose of Clenil® Modulite® | 0-12 hours
  Plasma AUC0-12h,ss for B17MP
Systemic exposure to B17MP (active metabolite of BDP) at steady state after repeated dose of Clenil® Modulite® | 0-12 hours
  Plasma Cmax,ss for B17MP

SECONDARY OUTCOMES:
evaluation of the pharmacokinetic profile of BDP | 0-12 hours
  AUC and Cmax for BDP
Vital signs assessment | from screening (week -1) to week 8
  Heart rate and Blood pressure assessment
haematology and blood chemistry assessment | at screening (week - 1) and week 8
  haematology and blood chemistry assessment
Number of patients with Adverse events | during the 11 weeks of study
  Adverse events
FEV1 predose assessment | from screening (week-1) to week 8
  FEV1 predose assessment as lung function parameter

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicine Evaluation Unit, Manchester, UK
Locations (1):
- Medicines Evaluation Unit, Wythenshawe Hospital, Manchester, United Kingdom

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2010-022615-19